CLINICAL TRIAL: NCT02990143
Title: The Effectiveness of Ologen® Collagen Matrix in Preventing Intraocular Pressure (IOP) Spikes After Ahmed Glaucoma Valve Surgery (AGV-FP7)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator left the Institution
Sponsor: The New York Eye & Ear Infirmary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13.33
Record Dates: First submitted 2016-12-06; First posted 2016-12-13 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — collagen-glycosaminoglycan copolymer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glaucoma Drainage implant no Ologen (No Intervention): The first group will use the routine technique for glaucoma drainage implant without placement of Ologen.
- Glaucoma Drainage implant with Ologen (Active Comparator): the second group will undergo the same procedure but will have the Ologen placed and secured over the plate of the AGV-FP7, under the conjunctiva, during the surgery.
  Interventions: Procedure: Ologen

INTERVENTIONS:
Procedure: Ologen — Ologen® CM,a biodegradable scaffold matrix, induces a regenerative non-scarring wound healing process without using anti-fibrotic agents.
  Arms: Glaucoma Drainage implant with Ologen

SUMMARY:
The purpose of this study is to investigate whether placing Ologen over the posterior plate of the Ahmed glaucoma drainage device during initial implantation will allow the formation of a thinner capsule, and decrease the incidence and/or the extent of IOP elevation during the postoperative period.

DETAILED DESCRIPTION:
Uncontrolled glaucoma may require surgical intervention. Glaucoma drainage implants such as AGV-FP7 are in wide use upon glaucoma and comprehensive surgeons. The success of aqueous shunt surgery depends on the formation and maintenance of a thin permeable capsule around the posterior plate of the aqueous shunt. Encapsulated bleb formation, where the capsule is thick and elevated, is a common cause of drainage failure in the early post-operative period. This finding is usually accompanied by elevated intraocular pressure (IOP), which requires additional intervention, often surgical and therefore reduces the success rate of the initial surgery.

Recently, a biodegradable porous collagen-glycosaminoglycan copolymer matrix implant (Ologen), has become available for glaucoma surgery. This device is constructed so as to minimize random growth of fibroblasts and instead to allow them to grow through the pores in the matrix. Ologen® CM,a biodegradable scaffold matrix, induces a regenerative non-scarring wound healing process without using anti-fibrotic agents.

This study is to investigate whether placing Ologen over the posterior plate of the Ahmed glaucoma drainage device during initial implantation will allow the formation of a thinner capsule, and decrease the incidence and/or the extent of IOP elevation during the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Uncontrolled treated glaucoma requiring AGV-FP7 surgery.
* Subject must be able and willing to cooperate with investigation plan.
* Subject must be able and willing to complete postoperative follow-up requirements
* Subject must be willing to sign informed consent form

Exclusion Criteria:

* Known allergic reaction to porcine collagen
* History of uveitis
* Corneal opacity or irregularity, preventing visualization of patency of tip of tube or accurate applanation
* History of scleral buckle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01-15 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
The Effectiveness of ologen® Collagen Matrix in preventing intraocular pressure (IOP) spikes after Ahmed Glaucoma Valve Surgery (AGV-FP7) | 1 year
  Ologen over the posterior plate of the Ahmed glaucoma drainage device during initial implantation will allow the formation of a thinner capsule, and decrease the incidence and/or the extent of IOP elevation during the postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Noga Harizman, MD, Principal Investigator — NY Eye Ear
Locations (1):
- New York Eye and Ear Infirmary, New York, New York, United States